CLINICAL TRIAL: NCT01330537
Title: Exploring the Visual Sensitivity for Topological Properties in Newborn Infants
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Sarina Hui-Lin Chien, Assistant Professor, China Medical University, China
Other Study IDs: DMR100-IRB-019
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Visual Sensitivity in Newborns
Keywords: perceptual development; topological perception theory; familiarization/novelty preference method; Discriminate a disk and a ring (topologically different),; Discriminate a disk and a triangle (geometrically different); Detect a change in the number of holes; Detect the size of the hole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The topological perception theory proposed a precise description for how one organizes the visual world that eliminates the vagueness of subjective phenomenology. In addition, the topological theory challenges the dominant computational view on the part-to-whole hierarchy of visual information processing. Lines of evidence from adult psychophysics, brain imaging data, and even honeybee's behavior have supported the notion that the global topological properties are the very primitives of visual representation. However, the question of how the sensitivity to topological properties originates during development has not been explored much. In a previous study, the investigators found that 2- to 6 month old infants could reliably discriminate stimuli based on topological differences, but failed to do so based on geometric differences. Using familiarization/novelty preference procedure, the present study intends to explore the visual sensitivity for topological properties in newborn infants. Experiment 1 focuses on whether neonates can discriminate a disk (no hole) and a ring (with a hole) that are topologically different, and/or a disk (no hole) and a triangle (no hole) that are geometrically different. Experiment 2 focuses on whether neonates can detect a change in the number of holes and/or the size of the hole. If newborn infants are only sensitive to topological properties and not to geometric properties, this will be a strong proof for the claim that topological property is the very "primitive" visual representation at empirical as well as theoretical level.

ELIGIBILITY:
Inclusion Criteria:

* full-term and healthy newborns

Exclusion Criteria:

* Eye illnesses or other physical problems

Ages: 3 Hours to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: full-term and healthy newborns
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Hui-Lin Chien, PhD, Principal Investigator — Graduate Institute of Neural and Cognitive Sciences, China Medical University, Taiwan; Bai-Horng Su, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taiwan